CLINICAL TRIAL: NCT00655122
Title: Double-Blind, Placebo-Controlled, Pilot Study, In Medical Patients With Prophylaxis Of Venous Thromboembolism in Primary Care
Brief Title: Prophylaxis In Venous Thromboembolism In Primary Care, A Pilot Study
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: See Detailed Description.
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: FGMAEI-0042-046; A6301036
Record Dates: First submitted 2008-04-04; First posted 2008-04-09 (Estimated); Last update posted 2008-09-29 (Estimated); Status verified 2008-09

CONDITIONS: Thromboembolism; Deep Vein Thrombosis; Dalteparin
MeSH Terms: conditions — Thromboembolism; Venous Thrombosis | interventions — Dalteparin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dalteparin sodium (Active Comparator)
  Interventions: Drug: Dalteparin sodium
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dalteparin sodium — Dalteparin sodium was administered at a daily dosage of 5,000 UI anti-Xa by subcutaneous route. The treatment duration was 7 days in a single daily injection throughout the bedridden period.
  Arms: Dalteparin sodium
Drug: Placebo — Placebo was administered with a daily injection of 0.2 mL by subcutaneous route. The treatment duration was 7 days in a single daily injection throughout the bedridden period.
  Arms: Placebo

SUMMARY:
The primary objective was to study the clinical benefit with dalteparin sodium in thromboprophylaxis in primary care medical subjects. The secondary objective was a pharmacoeconomic evaluation of hromboprophylaxis with dalteparin sodium in primary care medical subjects.

DETAILED DESCRIPTION:
The study was prematurely terminated on December 9, 2003. The reason for the early termination was not related to a safety or efficacy issue. It was related to the difficulty in recruiting patients.

ELIGIBILITY:
Inclusion Criteria:

* Age > 65 years
* Confinement to bed for more than 3 days, due to:
* Heart failure
* Exacerbated chronic obstructive pulmonary disease
* Acute rheumatic involvement
* Written informed consent

Exclusion Criteria:

1. Cancer
2. Anticoagulant treatment in the previous 3 months
3. Stroke or major surgery in the previous 3 months
4. Systolic pressure >200 mmHg or diastolic pressure >120 mmHg
5. Known chronic hepatopathy
6. Active hemorrhage in any site in the previous 3 months
7. Active peptic ulcer
8. Bacterial endocarditis
9. Conditions that can increase the risk of hemorrhage
10. Known coagulation disorders
11. Hypersensitivity to heparin or HIT
12. Life expectancy of less than 3 months
13. Previous confinement to bed during more than 3 days

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 8 (Actual)
Dates: Start 2003-04; Study Completion 2003-12 (Actual)

PRIMARY OUTCOMES:
Incidence of the endpoint made up of objectively demonstrated deep vein thrombosis (DVT), pulmonary embolism (PE) diagnosed by objective tests or death at the end of the follow-up period, 1 month after the end of the bedridden period. | 1 month

SECONDARY OUTCOMES:
Incidence of symptomatic deep vein thrombosis (DVT), symptomatic pulmonary embolism (PE) and tolerability at the end of the follow-up period. | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (4):
- Spain (4):
  - Pfizer Investigational Site, León
  - Pfizer Investigational Site, Madrid
  - Pfizer Investigational Site, Parla
  - Pfizer Investigational Site, Torremolinos

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=FGMAEI-0042-046&StudyName=Prophylaxis%20In%20Venous%20Thromboembolism%20In%20Primary%20Care%2C%20A%20Pilot%20Study